CLINICAL TRIAL: NCT04335890
Title: Phase I Vaccination Trial in Metastatic Uveal Melanoma Using IKKb-matured Dendritic Cells Loaded With Autologous Tumor-RNA + RNA Coding for Defined Antigens and Driver Mutations
Brief Title: IKKb-matured, RNA-loaded Dendritic Cells for Metastasised Uveal Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hasumi International Research Foundation (Other)
Responsible Party: Principal Investigator, Beatrice Schuler-Thurner, Ph.D, PD Dr. Beatrice Schuler-Thurner, University Hospital Erlangen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DERMA-ER-DC 09
Record Dates: First submitted 2020-04-01; First posted 2020-04-07 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Melanoma, Uveal Metastatic
Keywords: local treatment not sufficient; systemic treatment indicated
MeSH Terms: conditions — Melanoma | interventions — Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DC IKKb (Experimental): Vaccination with IKKb matured RNA loaded Dendritic Cells
  Interventions: Biological: Vaccination with IKKb matured Dendritic Cells

INTERVENTIONS:
Biological: Vaccination with IKKb matured Dendritic Cells — IKKb matured autologous monocyte derived dendritic cells loaded with RNAs; intravenous Infusion with a dose escalation starting with 7.5 mio Dendritic Cells for the first vaccination up to 30 mio cells per vaccination
  Other Names: Dendritic Cell vaccine

SUMMARY:
A Phase I vaccination trial in patients suffering from recently diagnosed metastatic uveal melanoma not cureable with local therapy and needing systemic therapy. IKKb-matured Dendritic Cells loaded with autologous tumor-RNA + RNA coding for defined antigens and driver mutations will be added to a standard therapy chosen by the tumor board (either checkpoint blockade or chemotherapy).

DETAILED DESCRIPTION:
Intravenous infusion of 7.5 to 30 mio DCIKKb at 9 vaccination time points (week 1, 3, 7, 13, 19, 25, 31, 37 and 42) and in intervals of 2, 4, and 6 intervals of 6 weeks) is scheduled; the first 4 patients will receive reduced doses for the first 4 vaccinations, namely 7.5 mio (1st and 2nd vaccination) and 15 mio (3rd and 4th vaccination) DC followed by the full dose of 30 mio for subsequent vaccinations. Patients number 5 to 8 will receive initially reduced doses of 15 mio (1st and 2nd vaccination) DC for the first 2 vaccinations, and the full dose of 30 mio for subsequent vaccinations. Patients number 8 to 12 will receive the full dose of 30 mio cells from vaccination 1 onwards provided that no major side effects occurred. Patients will be vaccinated in a staggered approach by selectively decelerating release of the vaccine.

DCIKKb = autologous, monocyte-derived DC that are matured with the standard cocktail (TNF-alpha, IL-1 beta, IL-6 and PGE2) and IKKb-RNA loaded by electroporation with 1) autologous PCR-amplified total tumor mRNA, 2) RNA coding for defined tumor associated antigens (TAA) namely gp100, tyrosinase, PRAME, MAGE-A3, IDO) and 3) RNA coding for driver mutations (GNAQ/GNA11Q209 or R183, or the less frequently occurring SF3B1R625, CYSLTR2L129Q or PLCB4D630) by electroporation; RNAs for selected TAAs are in stock and will be transfected into the DCs only if expressed in the individual tumor of a patient (shown by RNA sequencing of the tumor); RNAs for selected driver mutations are in stock and will be loaded into the DCs only if the respective mutation is found (proven by exome and RNA sequencing) in the individual tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable stage IV metastatic uveal melanoma as per AJCC staging system 2014, 7th edition (updated 2018) not curable with local therapy modalities
* WHO performance status of 0, 1 or 2
* age from 18 and ≤ 75 years
* negative pregnancy test
* signed informed consent

Exclusion Criteria:

* Major serious illness
* evidence for HIV-1, HIV-2, HTLV-1, HBV or HCV infection
* active autoimmune disease requiring immunosuppressive therapy
* splenectomy or radiation therapy of the spleen
* organ allografts
* pregnancy
* lactation
* psychiatric disorders
* severe organic brain syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety of DCIKKb | 1 year
  Assesment of side effects using the Common Toxicity Criteria (CTC v4.0)
Tolerability of DCIKKb | 1 year
  Assesment of Quality of life using Quality of life EORTC QLQ-C30, Version 2
Dose-limiting toxicities (DLTs) of DCIKKb | 1 year
  Assesment of side effects using the Common Toxicity Criteria (CTC v4.0)
Maximum tolerated dose (MTD) of DCIKKb | 1 year
  Assesment of side effects using the Common Toxicity Criteria (CTC v4.0)

SECONDARY OUTCOMES:
Prolongation of median overall survival | 2 years
  Assesment of survival
Prolongation of overall survival (OS) after 1 and 2 years | 2 years
  Assesment of survival
Induction of antigen specific CD8+ T cells and / or CD4+ T cells against TAA and mutated drivers | 2 years
  Assesment of immune responses

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Schuler-Thurner, MD, Principal Investigator — University Hospital Erlangen, Germany
Locations (1):
- University Hospital Erlangen Dept. of Dermatology, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pfeiffer IA, Hoyer S, Gerer KF, Voll RE, Knippertz I, Guckel E, Schuler G, Schaft N, Dorrie J. Triggering of NF-kappaB in cytokine-matured human DCs generates superior DCs for T-cell priming in cancer immunotherapy. Eur J Immunol. 2014 Nov;44(11):3413-28. doi: 10.1002/eji.201344417. Epub 2014 Sep 16. PMID 25100611
- [Result] Gerer KF, Erdmann M, Hadrup SR, Lyngaa R, Martin LM, Voll RE, Schuler-Thurner B, Schuler G, Schaft N, Hoyer S, Dorrie J. Preclinical evaluation of NF-kappaB-triggered dendritic cells expressing the viral oncogenic driver of Merkel cell carcinoma for therapeutic vaccination. Ther Adv Med Oncol. 2017 Jul;9(7):451-464. doi: 10.1177/1758834017712630. Epub 2017 Jun 13. PMID 28717398
- [Result] Schuler-Thurner B, Bartz-Schmidt KU, Bornfeld N, Cursiefen C, Fuisting B, Grisanti S, Heindl LM, Holbach L, Keseru M, Knorr H, Koch K, Kruse F, Meiller R, Metz C, Meyer-ter-Vehn T, Much M, Reinsberg M, Schliep S, Seitz B, Schuler G, Susskind D, Viestenz A, Wagenfeld L, Zeschnigk M. [Immunotherapy of uveal melanoma: vaccination against cancer. Multicenter adjuvant phase 3 vaccination study using dendritic cells laden with tumor RNA for large newly diagnosed uveal melanoma]. Ophthalmologe. 2015 Dec;112(12):1017-21. doi: 10.1007/s00347-015-0162-z. German. PMID 26602097
- [Derived] Koch EAT, Schaft N, Kummer M, Berking C, Schuler G, Hasumi K, Dorrie J, Schuler-Thurner B. A One-Armed Phase I Dose Escalation Trial Design: Personalized Vaccination with IKKbeta-Matured, RNA-Loaded Dendritic Cells for Metastatic Uveal Melanoma. Front Immunol. 2022 Feb 4;13:785231. doi: 10.3389/fimmu.2022.785231. eCollection 2022. PMID 35185883